CLINICAL TRIAL: NCT06436144
Title: A Single-Center, Prospective, Single-Arm, Observational Study Evaluating the Efficacy and Safety of Osimertinib Combined With Etoposide as First-Line Treatment in Patients With Osimertinib-Resistant or -Insensitive, Advanced EGFR-Mutant Non-Small Cell Lung Cancer
Brief Title: Osimertinib and Etoposide as First-Line Treatment in Osimertinib-Resistant Advanced EGFR-Mutant NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Yong He, Professor, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABC2024521
Record Dates: First submitted 2024-05-21; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Non Small Cell Lung Cancer; EGFR Gene Mutation; Non Small Cell Lung Cancer Stage IIIB; Non-small Cell Lung Cancer Stage IV
Keywords: Non Small Cell Lung Cancer; EGFR Gene Mutation; Primary drug resistance of oxitinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osimertinib Combined With Etoposide Soft Capsule (Experimental)
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Etoposide Soft Capsules Dosage：25mg/tablet, 2 tablets/time, taken continuously for 21 days, and stopped for one week. Osimertinib Dosage：80mg/tablet, 1 tablet/time, QD, taken for two cycles.
  Other Names: Etoposide Soft Capsules

SUMMARY:
Osimertinib, though a standard first-line treatment for EGFR-mutant advanced NSCLC, shows primary resistance in 10-30% of patients, leading to disease progression within 3-4 months. This resistance is linked to co-mutations in genes like TP53, RB1, and PIK3CA, among others. Studies indicate that Topo II inhibitor Etoposide (VP-16) can reduce cell survival, enhance DNA damage, and delay resistance in Osimertinib-resistant cells, suggesting a potential combination therapy to manage resistance.This study is a single-center, prospective, single-arm study evaluating the efficacy and safety of osimertinib combined with etoposide as a first-line treatment in patients with osimertinib-resistant or -insensitive advanced non-small cell lung cancer (NSCLC). The study focuses on patients with advanced NSCLC (stage IIIB or IV) with EGFR-sensitive mutations who developed slow resistance to osimertinib and for whom secondary biopsy after resistance did not identify any therapeutic targets.

DETAILED DESCRIPTION:
Although Osimertinib has become the standard first-line treatment choice for EGFRm advanced NSCLC, a subset of patients still do not benefit from first-line Osimertinib treatment. Some patients even experience disease progression at the initial stages of Osimertinib treatment. As early as 2010 and 2016, studies published in J Clin Oncol and Onco Targets Ther noted that approximately 10-30% of patients either do not respond to initial EGFR TKI treatment or experience disease control for less than 3 months despite carrying EGFR mutations (PMID: 19949011, 27382309). Furthermore, the FLAURA study on first-line Osimertinib treatment for EGFRm advanced NSCLC patients found that 3% of patients did not respond to Osimertinib, indicating potential primary resistance to Osimertinib (PMID: 29151359). This primary resistance is characterized by disease progression or stabilization within 3-4 months of EGFR TKI treatment, with no evidence of objective response during treatment (PMID: 27382309). Thus, primary resistance to third-generation EGFR-TKI Osimertinib significantly limits its clinical efficacy and presents a critical clinical challenge.

The mechanisms underlying primary resistance to Osimertinib are complex and not well understood, and research data are limited. Current evidence suggests that primary resistance to first-line Osimertinib in EGFRm advanced NSCLC patients may be related to concomitant co-mutations, such as atypical EGFR mutations and downstream/bypass pathway gene abnormalities (see Figure 1). Approximately 20-30% of EGFR mutation patients present with co-mutations at initial diagnosis, with common co-mutated genes including TP53 (54.6-64.6%), RB1 (9.6-10.33%), ERBB2 (8-11%), CTNNB1 (9.6%), PIK3CA (9-12.4%), and cell cycle-related genes like CDK4/CDK6/CCNE1, MET, KEAP1/NFE2L2/CUL3 axis, etc. These gene abnormalities can mediate primary resistance to EGFR-TKI therapy by activating EGFR bypass or downstream signaling pathways (PMID: 38382773, 37093192). A 2023 article in Targeted Oncology noted that TP53mutations, high AXL mRNA expression, and low BIM mRNA expression might be associated with poor response to Osimertinib (PMID: 37017806). Additionally, a case study published in Lung Cancer in 2023 reported that a patient with primary resistance to Osimertinib had simultaneous EGFR L858R and EGFR S645C mutations. After one month of Osimertinib treatment, there was no reduction in the right upper lobe nodule size, and CEA levels continued to rise. The patient continued with Osimertinib combined with anlotinib for four months, with no reduction in the primary tumor and persistently elevated CEA levels, indicating primary resistance to Osimertinib (PMID: 37842288). Other studies suggest that primary EGFR 20ins and BIM polymorphism deletion may mediate primary resistance to Osimertinib (PMID: 34669648). EGFR TKI primarily works by competitively binding to the ATP binding site, blocking EGFR phosphorylation and downstream signaling pathway activation, thus inducing tumor cell apoptosis. However, the crystal structure of EGFR 20ins does not affect the ATP binding pocket, preventing increased affinity between EGFR TKI and EGFR protein, leading to insensitivity and resistance to EGFR TKI therapy (PMID: 34301786). In patients with BIM gene abnormalities, compared to wild-type BIM, EGFR mutation patients with concurrent BIM deletion had lower ORR (28% vs 52.5%, P=0.026) and shorter PFS (8.3m vs 10.5m, P=0.031) following Osimertinib treatment (PMID: 34669648). Additionally, NSCLC patients with concurrent SCLC components or SCLC transformation may also exhibit primary resistance to Osimertinib (PMID: 29290257).Recent research has found that the DNA topoisomerase II (Topo II) inhibitor Etoposide (VP-16) synergistically reduces cell survival, enhances DNA damage and apoptosis induction in Osimertinib-resistant cells, inhibits the growth of Osimertinib-resistant tumors, and delays the emergence of acquired resistance to Osimertinib. Mechanistically, Osimertinib promotes proteasomal degradation mediated by fbxw7, leading to DNA damage and reduced Topo IIα levels in NSCLC cells; these effects are absent in Osimertinib-resistant cell lines with high Topo IIα levels. Elevated Topo IIα levels have also been detected in most EGFRm NSCLC tissues that recur after EGFR-TKI treatment. In sensitive EGFRm NSCLC cells, forced expression of ectopic TOP2A confers resistance to Osimertinib, whereas knocking down TOP2A in Osimertinib-resistant cell lines restores their response to Osimertinib-induced DNA damage and apoptosis. Overall, these findings reveal the important role of Topo IIα inhibition in mediating the therapeutic effects of Osimertinib on EGFRm NSCLC and provide a scientific rationale for targeting Topo II with Etoposide (VP-16) to manage Osimertinib-insensitive or primary-resistant cases (PMID: 38451729).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 79 years.
2. Locally advanced (stage IIIB) or metastatic (stage IV) EGFR-mutant NSCLC.
3. Harboring an EGFR sensitizing mutation (Exon 19 deletion or L858R).
4. Received at least two cycles of first-line osimertinib treatment, with a best response of stable disease or slow progression.
5. Life expectancy greater than 3 months.
6. At least one measurable tumor lesion meeting the following criteria:

1.No prior radiation therapy; 2.Measurable by chest CT or PET-CT, with a longest diameter ≥ 10 mm at baseline (short axis ≥ 15 mm for lymph nodes); 3.Amenable to accurate repeated measurements.

Exclusion Criteria:

1. Currently receiving or planning to receive other anti-cancer therapies.
2. Having contraindications to osimertinib or etoposide.
3. Harboring known targetable osimertinib resistance mechanisms.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Objective Remission Rate (ORR) as assessed by RECIST v1.1 | Within 1 month after treatment
  To evaluate the efficacy of osimertinib combined with etoposide as first-line treatment in patients with osimertinib-resistant or -insensitive, advanced EGFR-mutant non-small cell lung cancer. ORR will be defined as the proportion of patients achieving complete response (CR) or partial response (PR) according to RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Two-Year Overall Survival Rate | Up to 2 years after the start of treatment
  To observe the two-year overall survival rate of the treatment group receiving osimertinib combined with etoposide. OS will be measured from the start of treatment to the time of death from any cause.
One-Year Progression-Free Survival Rate | Up to 1 year after the start of treatment
  To observe the one-year tumor progression-free survival time in the treatment group receiving osimertinib combined with etoposide. PFS will be defined as the time from the start of treatment to the time of disease progression or death, whichever occurs first, as assessed by RECIST v1.1.
Disease Control Rate (DCR) within One Month | Within 1 month after treatment
  To observe the disease control rate in the treatment group receiving osimertinib combined with etoposide. DCR will be defined as the proportion of patients achieving complete response (CR), partial response (PR), or stable disease (SD) according to RECIST v1.1.
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | Within 1 month after treatment
  To observe the safety of osimertinib combined with etoposide in the treatment group. Safety will be assessed by the number of participants with treatment-related adverse events (AEs), graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

IPD SHARING:
Plan to Share IPD: Undecided